CLINICAL TRIAL: NCT00000331
Title: Buprenorphine/Naloxone Treatment for Opioid Dependence-Experiment II-3
Brief Title: Buprenorphine/Naloxone Treatment for Opioid Dependence-Experiment II-3 - 6
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-11160-6; R01DA011160 (NIH); R01-11160-6
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Heroin Dependence; Opioid-Related Disorders
Keywords: Heroin Dependence
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders | interventions — Drug Evaluation

ARMS (2):
- Test Drug (Experimental): Test drug to prevent heroine withdrawal
  Interventions: Drug: Test Drug
- Placebo Pill (Placebo Comparator): Placebo drug
  Interventions: Drug: Placebo Drug

INTERVENTIONS:
Drug: Test Drug
  Other Names: test drug o
  Arms: Test Drug
Drug: Placebo Drug
  Arms: Placebo Pill

SUMMARY:
The purpose of this study is to assess the abuse liability and examine the reinforcing effects of intravenous buprenorphine and buprenorphine/naloxone combinations in healthy, non-drug dependent volunteers.

DETAILED DESCRIPTION:
not available at this time

ELIGIBILITY:
Inclusion Criteria:

Individuals must be healthy, non-drug dependent volunteers, be at least 18 years of age, and have no prior history of drug or alcohol abuse or dependence. Subjects must have had some minimal experience with opioids (e.g. at least two prior exposures)

Exclusion Criteria:

Individuals with evidence of an active Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) Axis I psychiatric disorder (e.g. psychosis, manic-depressive illness, organic psychiatric disorders), significant medical illness (e.g., liver or cardiovascular disease) or pregnant female subjects are excluded from study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2002-12; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Observed withdrawal rating
Pupil diameter
Drug effect characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Amass, Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Health Sciences Center, Denver, Colorado, United States